CLINICAL TRIAL: NCT03506087
Title: Impact of Advance Care Planning Coaching for Patients With Chronic Kidney Disease
Brief Title: Advance Care Planning Coaching for Patients With Chronic Kidney Disease
Acronym: MY WAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Quality Insights (Unknown); Renal & Transplant Associates of New England (Unknown); Mountain Kidney and Hypertension Associates (Unknown); University of Pittsburgh (Other); Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Dale Lupu, Associate Research Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GW091617
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Chronic Kidney Diseases
Keywords: Advance Care Planning; Shared Decision Making
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to an intervention arm or an enhanced control arm. Participants in the intervention group will receive printed educational materials plus one or more ACP coaching sessions. Participants in the enhanced control arm will receive printed materials only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching (Experimental): Receives printed advance care planning (ACP) materials. Receives advance care planning coaching session. May receive followup coaching session, typically by telephone.
  Interventions: Behavioral: Advance care planning coaching session.; Behavioral: Printed advance care planning materials
- Enhanced Control (Active Comparator): Receives printed advance care planning materials only.
  Interventions: Behavioral: Printed advance care planning materials

INTERVENTIONS:
Behavioral: Advance care planning coaching session. — A 60-minute in-person coaching session. The advance care planning coach, trained in motivational interviewing, will use a flexible script and checklist to assess the participant's readiness to engage in advance care planning and guide the participant forward in the process, proceeding at the participant's pace. Some participants may complete advance directives while others will not get that far. Some participants may receive a follow-up session 2-4 weeks later. Typically this 20 to 30-minute conversation will be by phone, but it may be conducted at the clinic as indicated for the participant.
  Arms: Coaching
Behavioral: Printed advance care planning materials — Participants are provided with a folder containing an advance care planning guide developed by the Coalition for the Supportive Care of Kidney Patients for persons with Chronic Kidney Disease. The patient folder also contains the advance directive form used by the clinic that is appropriate to the state.

SUMMARY:
This project will develop and test a model intervention for Advance Care Planning (ACP) for patients with advanced chronic kidney disease (CKD) cared for in nephrology clinics that have the capacity to consult with or refer to palliative care. Specifically, we will compare the effectiveness of having a trained ACP coach meet in person with patients to discuss their goals and preferences vs. providing patients with a packet of material to review on their own and then discuss with their nephrologist at their initiation.

Hypothesis: In patients aged 55 or older with stage 3-5 Chronic Kidney Disease cared for in a CKD outpatient clinic, an advance care planning process that involves in-person meetings with a trained ACP coach will be more effective than providing patients with printed educational materials alone.

DETAILED DESCRIPTION:
BASELINE VISIT: After obtaining written informed consent, research staff will administer a baseline survey to assess ACP readiness as well as participant physical and emotional health. The participant will then be randomized to one of the study arms: intervention or control. Research staff will provide participants in both study arms with the advance care planning educational materials and instruct them that they are encouraged to discuss their thoughts and questions with the nephrologist, at their own initiation. Participants will be further encouraged to bring their advance directives (ADs) to the clinic to be scanned into the electronic health record (EHR) if they currently have ADs or complete them in the future.

ADVANCE CARE PLANNING COACHING SESSION (intervention arm only): Participants in the intervention arm will receive a 60-minute in-person coaching session. The advance care planning coach, trained in motivational interviewing, will use a flexible script and checklist to assess the participant's readiness to engage in advance care planning and guide the participant forward in the process, proceeding at the participant's pace. Some participants may complete advance directives while others will not get that far. The coach will document the clinical aspects of the discussion in the participant's medical chart according to clinic protocol and the research aspects in the participant tracking instruments. The ACP coach may arrange for one or more follow-up sessions as needed, typically conducted by telephone.

FOLLOW-UP ASSESSMENT SURVEY (both study arms): Approximately 14 weeks after the baseline visit, research staff will contact the participant to administer a follow-up assessment survey.

FOLLOW-UP CHART REVIEW: Approximately 16 weeks after the baseline visit, research staff will review the participant's medical chart to assess documentation of advance care planning activities, medical and health outcomes, and use of medical and palliative care services.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease (CKD) Stage 3-5
* Age 55 or older
* English speaking
* Patient at participating CKD clinic

Exclusion Criteria:

* Receiving dialysis
* Kidney transplant recipient
* Cognitively impaired or otherwise not competent to participate (as deemed by treating nephrologist and research staff)
* Participation contra-indicated for patient's health (as deemed by treating nephrologist)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Advance directive in EHR | 16 weeks after baseline
  Proportion of participants with advance directive or POLST/MOLST in EHR
ACP readiness score | 14 weeks after baseline
  Mean ACP readiness score at follow-up survey

SECONDARY OUTCOMES:
Medical decision maker documented in EHR | 16 weeks after baseline
  Proportion of participants with medical decision maker documented in EHR
ACP conversation with nephrologist documented in EHR | 16 weeks after baseline
  Proportion of participants with documentation in EHR of ACP conversation with nephrologist

CONTACTS AND LOCATIONS:
Overall Officials: Dale E Lupu, PhD, MPH, Principal Investigator — The George Washington University
Locations (4):
- United States (4):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Renal & Transplant Associates of New England, Springfield, Massachusetts
  - Mountain Kidney & Hypertension Associates, Asheville, North Carolina
  - University of Pittsburgh Medical Center Kidney Clinic, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lupu DE, Aldous A, Anderson E, Schell JO, Groninger H, Sherman MJ, Aiello JR, Simmens SJ. Advance Care Planning Coaching in CKD Clinics: A Pragmatic Randomized Clinical Trial. Am J Kidney Dis. 2022 May;79(5):699-708.e1. doi: 10.1053/j.ajkd.2021.08.019. Epub 2021 Oct 12. PMID 34648897